

Title: Takecab Tablets Special Drug Use Surveillance "Suppression of gastric or duodenal ulcer recurrence on non-steroidal anti-inflammatory drugs: Long-term use"

NCT Number: NCT03214198

Statistical analysis plan Approve Date: 09-NOV-2020

Certain information within this statistical analysis plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Patient identifiers within the text, tables, or figures or in by-patient data listings.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.

If needed, certain appendices that contain a large volume of personally identifiable information or company confidential information may be removed in their entirety if it is considered that they do not add substantially to the interpretation of the data (eg, appendix of investigator's curriculum vitae).

Note; This document was translated into English as the language on original version was Japanese.

# Statistical Analysis Plan

Takeda Pharmaceutical Company Limited

Takeda Pharmaceutical Company Limited Property of Takeda. For non-co

Version 1: Prepared on November 9, 2020

## Table of contents

| L | ist of | term | s/abbreviations | 3 |
|---|---|---|---|---|
| A | nalysi | is set | t | 5 |
| Ir | nporta | ant ic | dentified risks, important potential risks, and important missing information | 6 |
| Η | andlii | ng of | TIME WINDOW | 8 |
| H | andlir | ng of | f others | 9 |
| 1 | Nun | nber | of medical institutions, number of patients enrolled, and patient disposition | 10 |
| | 1.1 | Bre | akdown of patients (figure of patient disposition) | 210 |
| 2 | Pati | ent d | akdown of patients (figure of patient disposition)lemographics | . 12 |
| | 2.1 | Pati | ent demographics | . 12 |
| 3 | Trea | atme | nt details and concomitant drug. | 13 |
| | 3.1 | Stat | tus of treatment with Takecab Tablets | 13 |
| | 3.2 | Stat | tus of NSAID therapy | . 13 |
| | 3.3 | Con | ncomitant drug (excluding NSAIDs) | . 13 |
| 4 | Tab | ulate | d analysis on safety results | . 15 |
| | 4.1 | Inci | idence of AE and ADR/infection | . 15 |
| | 4. | 1.1 | tus of NSAID therapy accomitant drug (excluding NSAIDs) ad analysis on safety results idence of AE and ADR/infection Incidence of AE Incidence of ADR/infection | . 15 |
| | 4. | 1.2 | Incidence of ADR/infection | 16 |
| | | 1.3 | | |
| | | | identified risks, important potential risks, and important missing information | 17 |
| | 4.2 | Inci | dence of AE and ADR/infection in patients excluded from safety evaluation | 18 |
| | 4. | 2.1 | Incidence of AE | . 18 |
| | 4. | 2.2 | Incidence of ADR/infection | |
| | 4.3 | Inci | dence of AE and ADR/infection by seriousness, time of onset, and outcome | 20 |
| | | 3.1 | | |
| | 4. | 3.2 | | |
| | 4.4 | Inci | dence of ADR/infection by factor of patient demographics and treatment details | 22 |
| | 4. | 4.1 | Incidence of ADR/infection by factor of patient demographics and treatment details | 22 |
| | 4 | 4.2 | Incidence of ADR/infection by sex | |
| . ( | ¥4. | 4.3 | Incidence of ADR/infection by age subgroup | |
| 1 | 4. | 4.4 | Incidence of ADR/infection by purpose of NSAID therapy | |
| | 4. | 4.5 | Incidence of ADR/infection by presence/absence of complication | |
| | 4. | 4.6 | Incidence of ADR/infection by presence/absence of renal disease | |
| | | 4.7 | Incidence of ADR/infection by presence/absence of hepatic disease | |
| | | 4.8 | Incidence of ADR/infection by BMI subgroup | |
| | | | Incidence of ADR/infection by type of long-term NSAIDs | 26 |

| NSAIDs) | 27 |
|---|---|
| 4.4.11 Change of liver function test value | 27 |
| 5. Tabulated analysis on efficacy results | 28 |
| 5.1 Development of gastric ulcer, duodenal ulcer, or hemorrhagic lesions in stomach or | 20 |
| duodenum | 28 |
| 5.2 Development of gastric ulcer duodenal ulcer or hemorrhagic lesions in stomach or | 20 |
| duodenum (count in each subgroup) | 028 |
| 6. Incidence of ADR infection in additional pharmacovigilance activities | 30 |
| 6.1 Incidence of ADR/infection in additional pharmacovigilance activities (Attachment | 50 |
| Form 12) | 30 |
| 7 Outline of patients in postmarketing surveillance etc | 31 |
| 7.1 Outline of patients in postmarketing surveillance, etc. (Attachment Form 16) | 31 |
| Revision history (version control) | 32 |
| 1000 | |
| SULL | |
| 14.0. | |
| OU, | |
| SO | |
| i di | |
| No. | |
| alli. | |
| 2011 | |
| ada. | |
| i alko | |
| ×40. | |
| elc, | |
| A.4.11 Change of liver function test value. 5 Tabulated analysis on efficacy results 5.1 Development of gastric ulcer, duodenal ulcer, or hemorrhagic lesions in stomach or duodenum 5.2 Development of gastric ulcer, duodenal ulcer, or hemorrhagic lesions in stomach or duodenum (count in each subgroup). 6 Incidence of ADR/infection in additional pharmacovigilance activities. 6.1 Incidence of ADR/infection in additional pharmacovigilance activities (Attachment Form 12). 7 Outline of patients in postmarketing surveillance, etc. 7.1 Outline of patients in postmarketing surveillance, etc. (Attachment Form 16) | |
| X. | |

#### List of terms/abbreviations

- The drug: Takecab Tablets
- reaction and infection". Adverse events other than those analysis plan, the term "ADR/infection" is used in the title, and the term "ADR, etc." is used in the text and tables.

  Serious adverse event:

  An editor
- - An adverse event which the surveillance investigator assessed as "serious". Events included in the MedDRA code list of Takeda Medially Significant AE List are handled as serious even if the surveillance investigator assessed as "non-serious".
- Causality "related" to Takecab Tablets: The causality of an event not assessed as "not related" to Takecab Tablets is handled as "related", and the causality of an event assessed as "not related" to Takecab Tablets is handled as "not related".
- Summary statistics: An inclusive term of number of patients, mean, standard deviation, maximum value, minimum value, and quartile.
- Treatment days: The day before Takecab Tablets is started is Day -1, and the day when Takecab Tablets is started is Day 1.
- Duration (days) of treatment with Takecab Tablets: Completion date of treatment with Takecab Tablets - start date of treatment with Takecab Tablets + 1 (excluding days without treatment)
  - For patients with "under treatment with Takecab Tablets 12 months after the start of treatment" entered on the survey form, the duration of treatment is handled as 365 days (excluding days without treatment).
- Duration (days) of NSAID therapy: Completion date of NSAID therapy start date of NSAID therapy + 1 (excluding days without treatment)
  - For patients with missing completion date of NSAID therapy or "under NSAID therapy at the completion of survey" entered on the survey form, the duration of therapy is handled as missing (unknown).
  - For other patients with "therapy started before the start of treatment with Takecab Tablets" described as the status of NSAIDs on the survey form, but with missing start date, the duration of therapy is calculated by imputing "start time of NSAID therapy" described as patient demographics (the first date of the month is the start date of therapy). If only the

month is missing, "January 1" is imputed as the start date of therapy. Otherwise (both the year and month are missing or "unknown"), the duration of therapy is handled as missing Terms of Use (unknown).

- Patients whose survey forms have not been collected: In patients enrolled in the survey, patients whose survey forms have not been collected.
- Patients whose survey forms have been collected: In patients enrolled in this survey, patients BMI (kg/m²): Calculated as Weight (kg)/Height (m)² (rounded to the first decimal place).

   Time of onset of AE (ca. AB)? whose survey forms have been collected.
- Time of onset of AE (or ADR, etc.): When onset date of an AE (or ADR, etc.) is unknown, the A mon. aset are the active of first date of the month is the onset date. However, when the year and month of the start of Takecab Tablets and the year and month of AE (or ADR, etc.) onset are the same, the time of

4

#### Analysis set

In this survey, two analysis sets of "safety analysis set" and "efficacy analysis set" will be set.

Tablets with no significant protocol violation and evaluable for safety". In the patients whose survey forms have been collected, those falling under the following categories are excluded from the analysis set.

• Takecab Tablets was not an analysis set. the applica

- Administration of Takecab Tablets prior to contract period [found later]
- Enrollment in this survey 15 days or later after prescription of Takecab Tablets [found later]
- · It is unknown whether any AE developed or not

#### Efficacy analysis set

In this statistical analysis plan, "efficacy analysis set" is defined as "patients treated with Takecab Tablets with no significant protocol violation and evaluable for efficacy". In the safety analysis set, patients falling under the following categories are excluded from the efficacy analysis set.

- Other than target disease [found later]
- Patient failing to meet all of the inclusion criteria
- Patient meeting any of the exclusion criteria
- Patient with no post-baseline efficacy data
- Topical non-steroidal anti-inflammatory drug (NSAID) therapy only A post-baseline examination/physical examination was not conducted or was conducted outside the time window to determine the "development of gastric ulcer, duodenal ulcer, or

#### Important identified risks, important potential risks, and important missing information

- Important identified risk: Not applicable
- Important potential risk
- ierms of Use Hepatic function disorder: An AE falling under SMQ code 20000006 (Drug related hepatic disorders - comprehensive search [SMQ] narrow) is handled as hepatic function disorder.
  - Fracture: An AE falling under any of the PT codes listed in Table 1 is handled as fracture.
  - Gastrointestinal infection with clostridium difficile: An AE falling under SMQ code 20000080 (Pseudomembranous colitis [SMQ] narrow) is handled as gastrointestinal infection with clostridium difficile.
  - Neuroendocrine tumour due to increased serum gastrin: An AE falling under SMQ code 20000090 (Malignancies [SMQ] narrow) is handled as neuroendocrine tumour due to increased serum gastrin.
- · Important missing information: Not applicable

| PT NAME | PT CODE | PTNAME | PT CODE |
|---|---|---|---|
| Acetabulum fracture | 10000397 | Ilium fracture | 10021343 |
| Ankle fracture | 10002544 | Impacted fracture | 10066386 |
| Atypical femur fracture | 10070884 | Jaw fracture | 10023149 |
| Atypical fracture | 10072395 | Limb fracture | 10074551 |
| Avulsion fracture | 10066184 | Lower limb fracture | 10061599 |
| Bone fissure | 10064210 | Lumbar vertebral fracture | 10049947 |
| Bone fragmentation | 10064211 | Maisonneuve fracture | 10081343 |
| Cervical vertebral fracture | 10049946 | Metaphyseal corner fracture | 10079667 |
| Chance fracture | 10073162 | Multiple fractures | 10028200 |
| Clavicle fracture | 10009245 | Open fracture | 10030527 |
| Comminuted fracture | 10052614 | Osteophyte fracture | 10080550 |
| Complicated fracture | 10010149 | Osteoporotic fracture | 10031290 |
| Compression fracture | 10010214 | Patella fracture | 10034122 |
| Craniofacial fracture | 10077603 | Pathological fracture | 10034156 |
| Cuboid syndrome | 10081921 | Pelvic fracture | 10061161 |
| Epiphyseal fracture | 10053962 | Radius fracture | 10037802 |

| Facial bones fracture | Femoral neck fracture 10016450 Sacroiliac fracture 10074362 Femur fracture 10016454 Scapula fracture 10039579 Fibula fracture 10016667 Skull fracture 10061365 Foot fracture 10016970 Skull fractured base 10040960 Forearm fracture 10016997 Spinal compression fracture 10041541 Fracture 10017076 Spinal fracture 10041569 Fracture blisters 10079423 Spinal fusion fracture 10074807 Fracture displacement 10053206 Stapes fusion fracture 10042015 Fracture malunion 10017085 Sternal fracture 10042015 Fracture of clavicle due to birth trauma 10017107 Subchondral insufficiency fracture 10079864 Fractured coccyx 10049164 Thoracic vertebral fracture 10049948 Fractured sacrum 10017308 Tibia fracture 100493827 Fractured skull depressed 10017310 Totus fracture 10046094 Greenstick fracture 10018720 Traumatic fracture 10049514 | Femoral neck fracture 10016450 Sacroiliac fracture 10074362 Femur fracture 10016454 Scapula fracture 10039579 Fibula fracture 10016667 Skull fracture 10061365 Foot fracture 10016970 Skull fractured base 10040960 Forearm fracture 10016997 Spinal compression fracture 10041541 fracture Fracture 10017076 Spinal fracture 10041569 Fracture blisters 10079423 Spinal fusion fracture 10074807 Fracture displacement 10053206 Stapes fusion fracture 10081442 Fracture malunion 10017085 Sternal fracture 10042015 Fracture of clavicle due to birth trauma 10017108 Subchondral insufficiency fracture 10079864 insufficiency fracture Fractured occyx 10049164 Thoracic vertebral fracture 10049948 fracture Fractured sacrum 10017308 Tibia fracture 10049948 fracture Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10019114 Ulna fracture | Femoral neck fracture 10016450 Sacroiliac fracture 10074362 Femur fracture 10016454 Scapula fracture 10039579 Fibula fracture 10016667 Skull fracture 10061365 Foot fracture 10016970 Skull fracture dase 10040960 Forearm fracture 10016997 Spinal compression fracture 10041541 Fracture 10017076 Spinal fracture 10041569 Fracture blisters 10079423 Spinal fracture 10074807 Fracture displacement 10053206 Stapes fusion fracture 10081432 Fracture malunion 10017085 Sternal fracture 10042015 Fracture of clavicle due to birth trauma 10017107 Subchondral insufficiency fracture 100492212 Fractured coccyx 10049164 Thoracic vertebral fracture 10049948 Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Tous fracture 10066094 Greenstick fracture 10019114 Ulna fracture 10045375 Hi | PT NAME | PT CODE | PT NAME | PT CODE | |
|---|---|---|---|---|---|---|---|---|
| Forearm fracture | Forearm fracture | Forearm fracture | Forearm fracture | Facial bones fracture | 10016042 | Rib fracture | 10039117 | |
| Forearm fracture 10016997 Spinal compression fracture 10041541 Fracture 10017076 Spinal fracture 10041569 Fracture blisters 10079423 Spinal fusion fracture 10074807 Fracture displacement 10053206 Stapes fusion fracture 10081432 Fracture malunion 10017085 Sternal fracture 10042015 Fracture nonunion 10017088 Stress fracture 10042212 Fracture of clavicle due to birth trauma 10017107 Subchondral insufficiency fracture 10079864 Fractured coccyx 10049164 Thoracic vertebral fracture 10049948 Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10048049 | Forearm fracture | Forearm fracture | Forearm fracture | Femoral neck fracture | 10016450 | Sacroiliac fracture | 10074362 | |
| Forearm fracture | Forearm fracture | Forearm fracture | Forearm fracture | Femur fracture | 10016454 | Scapula fracture | 10039579 | 13 |
| Forearm fracture | Forearm fracture 10016997 Spinal compression fracture 10041541 Fracture 10017076 Spinal fracture 10041569 Fracture blisters 10079423 Spinal fusion fracture 10074807 Fracture displacement 10053206 Stapes fusion fracture 10081442 Fracture malunion 10017085 Sternal fracture 10042015 Fracture nonunion 10017088 Stress fracture 10042212 Fracture of clavicle due to birth trauma 10017107 Subchondral insufficiency fracture 10079864 Fractured coccyx 10049164 Thoracic vertebral fracture 10049948 Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10048049 | Forearm fracture 10016997 Spinal compression fracture 10041541 Fracture 10017076 Spinal fracture 10041569 Fracture blisters 10079423 Spinal fusion fracture 10074807 Fracture displacement 10053206 Stapes fusion fracture 10081442 Fracture malunion 10017085 Sternal fracture 10042015 Fracture nonunion 10017088 Stress fracture 10042212 Fracture of clavicle due to birth trauma 10017107 Subchondral insufficiency fracture 10079864 Fractured coccyx 10049164 Thoracic vertebral fracture 10049948 Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10048049 | Forearm fracture 10016997 Spinal compression fracture 10041541 Fracture 10017076 Spinal fracture 10041569 Fracture blisters 10079423 Spinal fusion fracture 10074807 Fracture displacement 10053206 Stapes fusion fracture 10081442 Fracture malunion 10017085 Sternal fracture 10042015 Fracture nonunion 10017088 Stress fracture 10042212 Fracture of clavicle due to birth trauma 10017107 Subchondral insufficiency fracture 10079864 Fractured coccyx 10049164 Thoracic vertebral fracture 10049948 Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10048049 | Fibula fracture | 10016667 | Skull fracture | 10061365 | 50' |
| Fracture 10017076 Spinal fracture 10041569 | Fracture 10017076 Spinal fracture 10041569 | Fracture 10017076 Spinal fracture 10041569 | Fracture 10017076 Spinal fracture 10041569 | Foot fracture | 10016970 | Skull fractured base | 10040960 | Sillis |
| Fracture blisters 10079423 Spinal fusion fracture 10074807 Fracture displacement 10053206 Stapes fusion fracture 10081442 Fracture malunion 10017085 Sternal fracture 10042015 Fracture nonunion 10017088 Stress fracture 010042212 Fracture of clavicle due to birth trauma 10017107 Subchondral insufficiency fracture 10079864 Fractured coccyx 10049164 Thoracic vertebral fracture 10049948 Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10048049 Wrist fracture 10048049 | Fracture blisters 10079423 Spinal fusion fracture 10074807 Fracture displacement 10053206 Stapes fusion fracture 10081442 Fracture malunion 10017085 Sternal fracture 10042015 Fracture nonunion 10017088 Stress fracture 10042212 Fracture of clavicle due to birth trauma 10017107 Subchondral insufficiency fracture 10079864 Fractured coccyx 10049164 Thoracic vertebral fracture 10049948 Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Fracture blisters 10079423 Spinal fusion fracture 10074807 Fracture displacement 10053206 Stapes fusion fracture 10081442 Fracture malunion 10017085 Sternal fracture 10042015 Fracture nonunion 10017088 Stress fracture 10042212 Fracture of clavicle due to birth trauma 10017107 Subchondral insufficiency fracture 10079864 Fractured coccyx 10049164 Thoracic vertebral fracture 10049948 Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10048049 Wrist fracture 10048049 | Fracture blisters 10079423 Spinal fusion fracture 10074807 Fracture displacement 10053206 Stapes fusion fracture 10081442 Fracture malunion 10017085 Sternal fracture 10042015 Fracture nonunion 10017088 Stress fracture 10042212 Fracture of clavicle due to birth trauma 10017107 Subchondral insufficiency fracture 10079864 Fractured coccyx 10049164 Thoracic vertebral fracture 10049948 Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10048049 Wrist fracture 10048049 | Forearm fracture | 10016997 | | 10041541 | Xo. |
| Fracture displacement 10053206 Stapes fusion fracture 10081442 Fracture malunion 10017085 Sternal fracture 10042015 Fracture nonunion 10017088 Stress fracture 10042212 Fracture of clavicle due to birth trauma 10017107 Subchondral insufficiency fracture 10079864 Fractured coccyx 10049164 Thoracic vertebral fracture 10049948 Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10048049 Wrist fracture 10048049 | Fracture displacement 10053206 Stapes fusion fracture 10081442 Fracture malunion 10017085 Sternal fracture 10042015 Fracture nonunion 10017088 Stress fracture 10042212 Fracture of clavicle due to birth trauma 10017107 Subchondral insufficiency fracture 10079864 Fractured coccyx 10049164 Thoracic vertebral fracture 10049948 Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Fracture displacement 10053206 Stapes fusion fracture 10081442 Fracture malunion 10017085 Sternal fracture 10042015 Fracture nonunion 10017088 Stress fracture 10042212 Fracture of clavicle due to birth trauma 10017107 Subchondral insufficiency fracture 10079864 Fractured coccyx 10049164 Thoracic vertebral fracture 10049948 Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Fracture displacement 10053206 Stapes fusion fracture 10081442 Fracture malunion 10017085 Sternal fracture 10042015 Fracture nonunion 10017088 Stress fracture 10042212 Fracture of clavicle due to birth trauma 10017107 Subchondral insufficiency fracture 10079864 Fractured coccyx 10049164 Thoracic vertebral fracture 10049948 Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Fracture | 10017076 | Spinal fracture | 10041569 | |
| Fracture malunion 10017085 Sternal fracture 10042015 Fracture nonunion 10017088 Stress fracture 10042212 Fracture of clavicle due to birth trauma 10017107 Subchondral insufficiency fracture 10079864 Fractured coccyx 10049164 Thoracic vertebral fracture 10049948 Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10048049 Wrist fracture 10048049 | Fracture malunion 10017085 Sternal fracture 10042015 Fracture nonunion 10017088 Stress fracture 10042212 Fracture of clavicle due to birth trauma 10017107 Subchondral insufficiency fracture fractured coccyx 10049164 Thoracic vertebral fracture 10049948 fracture Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Fracture malunion 10017085 Sternal fracture 10042015 Fracture nonunion 10017088 Stress fracture 10042212 Fracture of clavicle due to birth trauma 10017107 Subchondral insufficiency fracture 10049864 insufficiency fracture Fractured coccyx 10049164 Thoracic vertebral fracture Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Fracture malunion 10017085 Sternal fracture 10042015 Fracture nonunion 10017088 Stress fracture 100042212 Fracture of clavicle due to birth trauma 10017107 Subchondral insufficiency fracture fractured coccyx 10049164 Thoracic vertebral fracture 10049948 fracture Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Fracture blisters | 10079423 | Spinal fusion fracture | 10074807 | |
| Fracture of clavicle due to birth trauma Fractured coccyx Fractured sacrum Fractured skull depressed Greenstick fracture 10017107 10017308 Fractured skull depressed 10017310 Fractured skull depressed 10018720 Fractured fracture 10049514 Hand fracture 10020100 Upper limb fracture 10048049 Fracture 10048049 Humerus fracture 10048049 | Fracture nonunion 10017088 Stress fracture 10042212 Fracture of clavicle due to birth trauma 10017107 Subchondral insufficiency fracture 10079864 Fractured coccyx 10049164 Thoracic vertebral fracture 10049948 Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Fracture nonunion 10017088 Stress fracture 10042212 Fracture of clavicle due to birth trauma 10017107 Subchondral insufficiency fracture 10079864 Fractured coccyx 10049164 Thoracic vertebral fracture 10049948 Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Fracture nonunion 10017088 Stress fracture 10042212 Fracture of clavicle due to birth trauma 10017107 Subchondral insufficiency fracture 10049948 Fractured coccyx 10049164 Thoracic vertebral fracture 10049948 Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Fracture displacement | 10053206 | Stapes fusion fracture | 10081442 | |
| Fracture of clavicle due to birth trauma Fractured coccyx 10049164 Fractured sacrum 10017308 Fractured skull depressed 10017310 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10020100 Upper limb fracture 10048049 Wrist fracture 10048049 | Fracture of clavicle due to birth trauma Fractured coccyx 10049164 Fractured sacrum Fractured sacrum 10017308 Tibia fracture 10049827 Fractured skull depressed 10017310 Torus fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10048049 Wrist fracture 10048049 | Fracture of clavicle due to birth trauma Fractured coccyx 10049164 Fractured sacrum Fractured sacrum 10017308 Tibia fracture 10049827 Fractured skull depressed 10017310 Torus fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10048049 Wrist fracture 10048049 | Fracture of clavicle due to birth trauma Fractured coccyx 10049164 Fractured sacrum Fractured skull depressed Greenstick fracture 10019114 Humerus fracture 10017107 Subchondral insufficiency fracture 10049948 Thoracic vertebral 10049948 Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10048049 | Fracture malunion | 10017085 | Sternal fracture | 10042015 | |
| birth trauma insufficiency fracture Fractured coccyx 10049164 Thoracic vertebral fracture Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | birth trauma insufficiency fracture Fractured coccyx 10049164 Thoracic vertebral fracture Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | birth trauma insufficiency fracture Fractured coccyx 10049164 Thoracic vertebral fracture Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | birth trauma insufficiency fracture Fractured coccyx 10049164 Thoracic vertebral fracture Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Fracture nonunion | 10017088 | Stress fracture | 10042212 | |
| Fractured coccyx 10049164 Thoracic vertebral fracture 10049948 Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Fractured coccyx 10049164 Thoracic vertebral fracture 10049948 Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Fractured coccyx 10049164 Thoracic vertebral fracture 10049948 Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Fractured coccyx 10049164 Thoracic vertebral fracture 10049948 Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | | 10017107 | Subchondral insufficiency fracture | 10079864 | |
| Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Fractured sacrum 10017308 Tibia fracture 10043827 Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | | 10049164 | Thoracic vertebral | 10049948 | |
| Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Fractured skull depressed 10017310 Torus fracture 10066094 Greenstick fracture 10018720 Traumatic fracture 10049514 Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Fractured sacrum | 10017308 | | 10043827 | |
| Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Hand fracture 10019114 Ulna fracture 10045375 Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Fractured skull depressed | 10017310 | 10. | 10066094 | |
| Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Hip fracture 10020100 Upper limb fracture 10061394 Humerus fracture 10020462 Wrist fracture 10048049 | Greenstick fracture | 10018720 | Traumatic fracture | 10049514 | |
| Humerus fracture 10020462 Wrist fracture 10048049 | Humerus fracture 10020462 Wrist fracture 10048049 | Humerus fracture 10020462 Wrist fracture 10048049 | Humerus fracture 10020462 Wrist fracture 10048049 | Hand fracture | 10019114 | Ulna fracture | 10045375 | |
| | | | | Hip fracture | 10020100 | Upper limb fracture | 10061394 | |
| N-COMMRe. | . For non-comme | oxeda. For non-comme | akedai. For non-comme | Humerus fracture | 10020462 | Wrist fracture | 10048049 | |
| | . For no. | Hedai. For no. | Kakeda: For no. | | 10020462 | Wrist fracture | 10048049 | |
| (akedia. | C.O. | | | | | | | |
| (akeda. | C.O. | | | , o | | | | |
| Kakeda. | | | | , o | | | | |

#### Handling of TIME WINDOW

Data of tests/observations/endpoints which are evaluable (i.e., data which are not missing and are

The time window will be adopted. If there are multiple standard day will be adopted. If the number of days from the standard day is the same or the standard day is not specified, data of the later date will be adopted. The difference from the standard day is determined based on the post-treatment days. day is not specified, data of the later date will be adopted. The difference from the standard day is determined based on the post-treatment days.

Laboratory tests (AST, ALT, γ-GTP, ALP, Total bilirubin, LDH, Serum gastrin)

| Assessment time | Standard day of conduct | Time window Post-treatment days |
|---|---|---|
| At the start of treatment | Post-treatment days: -1 | -8 to 1 |
| At the completion of survey | Post-treatment days: - | Sulpile 2 or more |

Development of gastric ulcer, duodenal ulcer, or hemorrhagic lesions in stomach or duodenum

| <u>L</u> | Development of gastric tileer, duodenat tileer, of neurormagic lesions in stomach of duodentin | | |
|---|---|---|---|
| | Assessment time | Standard day of conduct | Time window Post-treatment days |
| | At the completion of survey | Post-treatment days: - | 2 or more |
| | | ORM | |
| | " non" | | |
| | At the completion of survey | | |
| .< | sker. | | |
| io kis | | | |
| Drobe. | | | |

## Handling of others

Property of Takeda. For non-commercial use only and subject to the applicable Tames of Use

#### 1 Number of medical institutions, number of patients enrolled, and patient disposition

#### Breakdown of patients (figure of patient disposition)

Analysis All patients enrolled in this survey (patients enrolled)

population:

Patients enrolled Analysis items:

Number of medical institutions

Patients whose survey forms have not

been collected

Patients whose survey forms have been

collected

Patients excluded from safety

evaluation\*

Reason of exclusion (multiple

counts)

the applicable Terms of Use ts not [Takecab Tablets not administered,

Administration prior to contract

period [found later], Enrollment 15

days or later after prescription of

Takecab Tablets [found later],

Unknown whether any AE developed or not]

Patients targeted for safety evaluation\*

Patients excluded from efficacy

evaluation\*

Reason of exclusion (multiple

[Other than target disease [found later],

Patient failing to meet all of the

inclusion criteria, Patient meeting

any of the exclusion criteria, Patient

with no post-baseline efficacy data,

Topical non-steroidal anti-

inflammatory drug (NSAID) therapy

only

Patients targeted for efficacy

Analysis method: Following analysis will be conducted for the above analysis items, and a figure

of patient disposition will be prepared.

Property of Takeda. For non-courts The number of medical institutions will also be calculated concerning patients enrolled in the survey. If patients are enrolled in more than one department in one medical institution, the number of the medical institution is counted as one.

10

Number of patients excluded from safety evaluation and efficacy evaluation are

- andicates seri. Takeda, for nonconfinercial use only and subject to the applicable of the property of takeda, for nonconfinercial use only and subject to the applicable of the property of takeda.

#### 2 Patient demographics

#### Patient demographics 2.1

Analysis Safety analysis set

population:

Analysis items: Sex

Age (year)

Previous medical history

(multiple counts)

[Min<= - <65, ≥65<= - <75, ≥75<= - <=Max]
[Gastric ulcer, Duodenal ulcer] [Rheumatoid arthritis, Osteoarthritis, Others] Purpose of NSAID therapy

(multiple counts)

[Outpatient, Inpatient] Inpatient/outpatient

classification

Existence of hypersensitivity [Yes or No or Unknown]

predisposition

Existence of complication

Height (cm) Weight (kg)

BMI  $(kg/m^2)$ 

25.0<= - <= Max]

Existence of H. pylori infection [Positive or Negative or Unknown]

[Non-smoker, Current smoker, Ex-smoker, Smoking history

Unknown]

Drinking history [Yes or No or Unknown] [Yes or No or Unknown]

Existence of stress, a risk factor

for developing gastric or

duodenal ulcer

Existence of acid-suppressant [Yes or No or Unknown]

therapy before the start of treatment with Takecab Tablets to prevent recurrent gastric or

duodenal ulcer

Breakdown of drugs in patients [Lansoprazole, Omeprazole, Rabeprazole,

with "Yes" Esomeprazole, H<sub>2</sub>-blocker]

Property of Takeda. For Analysis method: Following analysis will be conducted for the above analysis items.

(1) Frequency counts of countable data, and summary statistics of quantitative data

#### Treatment details and concomitant drug

#### Status of treatment with Takecab Tablets

Analysis Safety analysis set

population:

Initial daily dose of Takecab [10 mg, Others] Analysis items:

**Tablets** 

Duration (days) of treatment

[1<= -<=84, 85<= -<=168, 169<= -<=Max]

with Takecab Tablets

Reasons for discontinuation

[Incidence of AE, No patient visit due to reasons

of treatment with Takecab

such as changing hospital, Pregnancy,

**Tablets** 

Development of gastric ulcer/duodenal ulcer/hemorrhagic lesions in stomach or

duodenum, Discontinuation of NSAID

therapy, Others]

Analysis method: Following analysis will be conducted for the above analysis items.

(1) Frequency counts of countable data, and summary statistics of quantitative

data

#### Status of NSAID therapy 3.2

Analysis Safety analysis set

population:

Type of long-term NSAIDs Analysis items:

[COX-2 selective inhibitors, Others]

(at the initial dose)

Purpose of treatment with

Takecab Tablets after the

completion of NSAID

therapy

[Treatment of complication, Development of

gastric ulcer/duodenal ulcer/hemorrhagic

lesions in stomach or duodenum, Development of new gastrointestinal disease not mentioned

above after treatment with Takecab Tablets,

Others (e.g., prophylactic treatment)]

Analysis method: Following analysis will be conducted for the above analysis items.

(1) Frequency counts of countable data, and summary statistics of quantitative

data

#### Concomitant drug (excluding NSAIDs)

Analysis Safety analysis set

population:

Analysis items: Existence of concomitant drug (excluding [Yes or No]

NSAIDs)

Type of concomitant drug (excluding

NSAIDs)

properly of Takeda. For non-confinercial use only and subject to the applicable Tames of Use Analysis method: Following analysis will be conducted for the above analysis items. Concomitant

14

#### 4 Tabulated analysis on safety results

#### Incidence of AE and ADR/infection

#### 4.1.1 Incidence of AE

Analysis

Safety analysis set

population:

Analysis items:

Adverse event

Analysis method: Following analysis will be conducted for the above analysis items.

- Number of patients with AEs (1)
- (2)Number of incidence of AEs
- Percentage of patients with AEs (3)
- (4)Classification of AE

applicable Terms of Use The methods to count data for individual analyses are shown below.

[Number of patients with AEs]

Number of patients who experienced AEs.

[Number of incidence of AEs]

Number of AEs which developed. When an AE developed multiple times in a single patient, total number of events will be counted.

[Percentage of patients with AEs]

To be calculated with number of patients with AEs/number of patients targeted for safety evaluation x 100.

[Classification of AE]

AEs will be coded to MedDRA/J terms. AEs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).

SOC will be presented with number and percentage of patients with AEs in the internationally agreed order of SOC. When multiple events coded to terms in an identical SOC developed in a single patient, one patient will be counted for the SOC.

Property of Takedai. For non PT will be presented with number and percentage of patients with AEs in ascending order of PT codes. When multiple events coded to terms in an identical PT developed in a single patient, one patient will be counted for the PT.

#### 4.1.2 Incidence of ADR/infection

Analysis Safety analysis set

population:

Analysis items:

Analysis method: Following analysis will be conducted for the above analysis items.

[Percentage of patients with ADRs, etc.]

To be calculated with number of patients with ADRs, etc./number of patients targeted for safety evaluation x 100.

[Classification of ADRs, etc.]

- ADRs, etc. will be coded to MedDRA/J terms. AEs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and percentage of patients with ADRs, etc. in the internationally agreed order of SOC. When multiple events coded to terms in an identical SOC developed in a single patient, one patient will be counted for the SOC.
- Property of Takedai. For non PT will be presented with number and percentage of patients with ADRs, etc. in ascending order of PT codes. When multiple events coded to terms in an identical PT developed in a single patient, one patient will be counted for the PT.

# 4.1.3 Incidence of AE and ADR/infection falling under the categories of important identified risks, important potential risks, and important missing information

#### 4.1.3.1 Incidence of AEs falling under the category of safety specification (count by risk)

Analysis Safety analysis set

population:

Analysis items: AEs, etc. falling under the category of safety specification (described as

important identified risks, important potential risks, and important missing

information)

Subgroup items: Seriousness

[Serious, Non-serious]

Analysis method: Following analyses will be conducted for the above analysis items in each

subgroup by risk. The risks are important identified risks, important potential

risks, and as defined in important missing information.

[Classification of AE]

 AEs will be coded to MedDRA/J terms. AEs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).

- SOC will be presented with number and proportion of patients with AEs in
  the internationally agreed order of SOC. When multiple events coded to
  terms in an identical SOC developed in a single patient, one patient will be
  counted for the SOC. However, when the multiple events differ in
  seriousness, one patient will be counted as both serious and non-serious.
- PT will be presented with number and proportion of patients with AEs in
  ascending order of PT codes. When multiple events coded to terms in an
  identical PT developed in a single patient, one patient will be counted for
  the PT. However, when the multiple events differ in seriousness, one patient
  will be counted as both serious and non-serious.

# 4.1.3.2 Incidence ADRs/infections falling under the category of safety specification (count by risk)

Analysis

Safety analysis set

population:

Analysis items: ADRs, etc. falling under the category of safety specification (described as

important identified risks, important potential risks, and important missing

information)

Subgroup items: Seriousness

[Serious, Non-serious]

Analysis method: Following analyses will be conducted for the above analysis items in each subgroup by risk. The risks are important identified risks, important potential risks, and as defined in important missing information.

[Classification of ADRs, etc.]

- ADRs, etc. will be coded to MedDRA/J terms. ADRs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and proportion of patients with ADRs, etc. in the internationally agreed order of SOC. When multiple events coded to terms in an identical SOC developed in a single patient, one patient will be counted for the SOC. However, when the multiple events differ in seriousness, one patient will be counted as both serious and non-serious.
- PT will be presented with number and proportion of patients with ADRs, etc. in ascending order of PT codes. When multiple events coded to terms in an identical PT developed in a single patient, one patient will be counted for the PT. However, when the multiple events differ in seriousness, one patient will be counted as both serious and non-serious.

## Incidence of AE and ADR/infection in patients excluded from safety evaluation

#### 4.2.1 Incidence of AE

Patients excluded from safety analysis set Analysis

population:

Analysis items: Adverse event

Analysis method: Following analysis will be conducted for the above analysis items. Property of Takeda. For

- Number of patients with AEs
- (2)Number of incidence of AEs
- (3)Percentage of patients with AEs
- Classification of AE (4)

The methods to count data for individual analyses are shown below.

[Number of patients with AEs]

Number of patients who experienced AEs.

[Number of incidence of AEs]

Number of AEs which developed. When an AE developed multiple times in a single patient, total number of events will be counted.

[Percentage of patients with AEs]

 To be calculated with number of patients with AEs/number of patients targeted for safety evaluation x 100.

[Classification of AE]

- AEs will be coded to MedDRA/J terms. AEs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and percentage of patients with AEs in
  the internationally agreed order of SOC. When multiple events coded to
  terms in an identical SOC developed in a single patient, one patient will be
  counted for the SOC.
- PT will be presented with number and percentage of patients with AEs in ascending order of PT codes. When multiple events coded to terms in an identical PT developed in a single patient, one patient will be counted for the PT.

#### 4.2.2 Incidence of ADR/infection

Analysis Patients excluded from safety analysis set

population:

Property of Takedai. For

Analysis items: ADRs, etc.

Analysis method: Following analysis will be conducted for the above analysis items.

- (1) Number of patients with ADRs, etc.
- (2) Number of incidence of ADRs, etc.
- (3) Percentage of patients with ADRs, etc.
- (4) Classification of ADRs, etc.

The methods to count data for individual analyses are shown below.

[Number of patients with ADRs, etc.]

Number of patients who experienced ADRs, etc.

[Number of incidence of ADRs, etc.]

Number of ADRs, etc. which developed. When an ADR, etc. developed
multiple times in a single patient, total number of events will be counted.

[Percentage of patients with ADRs, etc.]

 To be calculated with number of patients with ADRs, etc./number of patients targeted for safety evaluation x 100.

[Classification of ADRs, etc.]

 ADRs, etc. will be coded to MedDRA/J terms. AEs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).

- SOC will be presented with number and percentage of patients with ADRs, etc. in the internationally agreed order of SOC. When multiple events coded to terms in an identical SOC developed in a single patient, one patient will be counted for the SOC.
- PT will be presented with number and percentage of patients with ADRs,
   etc. in ascending order of PT codes. When multiple events coded to terms in an identical PT developed in a single patient, one patient will be counted for the PT.

#### 4.3 Incidence of AE and ADR/infection by seriousness, time of onset, and outcome

#### 4.3.1 Incidence of AE by seriousness, time of onset, and outcome

Analysis Safety analysis set

population:

Property of Takeda. For

Analysis items: Adverse event

Subgroup items: Seriousness [Serious, Non-serious]

Time of onset (days) [1<= - <=84, 85<= - <=168, 169<= - <=Max, Unknown]

Outcome [Resolved, Resolving, Not resolved, Resolved with

sequelae, Death (due to the relevant event), Unknown]

Analysis method: Following analysis will be conducted for the above analysis items in each subgroup.

- (1) Number of patients with AEs
- (2) Number of incidence of AEs
- (3) Percentage of patients with AEs
- 4) Classification of AE

The methods to count data for individual analyses are shown below.

[Number of patients with AEs]

Number of patients who experienced AEs.

[Number of incidence of AEs]

 Number of AEs which developed. When an AE developed multiple times in a single patient, total number of events will be counted.

[Percentage of patients with AEs]

 To be calculated with number of patients with AEs/number of patients targeted for safety evaluation x 100.

[Classification of AE]

- AEs will be coded to MedDRA/J terms. AEs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and percentage of patients with AEs in
  the internationally agreed order of SOC. When multiple events coded to
  terms in an identical SOC developed in a single patient, one patient will be
  counted for the SOC. However, in an identical SOC, one event is adopted
  according to the priority order specified at the foot note.
- PT will be presented with number and percentage of patients with AEs in
  ascending order of PT codes. When multiple events coded to terms in an
  identical PT developed in a single patient, one patient will be counted for
  the PT. However, for an identical PT, one event is adopted according to the
  following order of priority.

Seriousness: Serious → Non-serious

Time of onset: The event which developed earliest after Takecab Tablets was started

Outcome: Death (due to the relevant event)  $\rightarrow$  Resolved with sequelae  $\rightarrow$  Not resolved  $\rightarrow$  Resolving  $\rightarrow$  Resolved  $\rightarrow$  Unknown

#### 4.3.2 Incidence of ADR/infection by seriousness, time of onset, and outcome

Analysis Safety analysis set

population:

Analysis items: ADRs, etc

Subgroup items: Seriousness [Serious, Non-serious]

Time of onset (days) [1 <= - <= 84, 85 <= - <= 168, 169 <= - <= Max,

Unknown]

Outcome [Resolved, Resolving, Not resolved, Resolved with

sequelae, Death (due to the relevant event),

Unknown]

Analysis method: Following analysis will be conducted for the above analysis items in each subgroup.

- (1) Number of patients with ADRs, etc.
- (2) Number of incidence of ADRs, etc.
- (3) Percentage of patients with ADRs, etc.
- (4) Classification of ADRs, etc.

The methods to count data for individual analyses are shown below.

#### [Number of patients with ADRs, etc.]

Number of patients who experienced ADRs, etc.

[Number of incidence of ADRs, etc.]

Number of ADRs, etc. which developed. When an ADR, etc. developed
multiple times in a single patient, total number of events will be counted.

[Percentage of patients with ADRs, etc.]

 To be calculated with number of patients with ADRs, etc./number of patients targeted for safety evaluation x 100.

[Classification of ADRs, etc.]

- ADRs, etc. will be coded to MedDRA/J terms. ADRs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and percentage of patients with ADRs, etc. in the internationally agreed order of SOC. When multiple events coded to terms in an identical SOC developed in a single patient, one patient will be counted for the SOC. However, in an identical SOC, one event is adopted according to the priority order specified at the foot note.
- PT will be presented with number and percentage of patients with ADRs, etc. in ascending order of PT codes. When multiple events coded to terms in an identical PT developed in a single patient, one patient will be counted for the PT. However, for an identical PT, one event is adopted according to the following order of priority.

Seriousness: Serious → Non-serious

Time of onset: The event which developed earliest after Takecab Tablets was started

Outcome: Death (due to the relevant event)  $\rightarrow$  Resolved with sequelae  $\rightarrow$  Not resolved  $\rightarrow$  Resolving  $\rightarrow$  Resolved  $\rightarrow$  Unknown

4.4 Incidence of ADR/infection by factor of patient demographics and treatment details

4.4.1 Incidence of ADR/infection by factor of patient demographics and treatment details

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Sex [Male, Female]

Age (year) [Min<= - <65, 65<= - <75,

 $75 \le - \le Max$ 

[Rheumatoid arthritis, Osteoarthritis, Purpose of NSAID therapy (multiple

counts)

[Yes or No]

[Min<= - <18.5, 18.5<= - <25.0,
25.0<= - <=Max]

[COX-2 inhibitors,
Others]

Yes or No]

Palent Service S Existence of complication Existence of renal disease Existence of hepatic disease

BMI (kg/m<sup>2</sup>)

Type of long-term NSAIDs (at the

initial dose) Existence of concomitant drug

(excluding NSAIDs)

Analysis method: Following analysis will be conducted for the above analysis items in each subgroup, and chi-square test will be conducted as reference (excluding items

falling under the category of multiple counts)

- Number of patients with ADRs, etc. (1)
- Percentage of patients with ADRs, etc. and its 95% confidence interval (2)(two-sided)

The methods to count data for individual analyses are shown below.

[Number of patients with ADRs, etc.]

Number of patients who experienced ADRs, etc.

[Percentage of patients with ADRs, etc.]

To be calculated with number of patients with ADRs, etc./number of patients targeted for safety evaluation x 100.

## 4.4.2 Incidence of ADR/infection by sex

Safety analysis set Analysis

population:

Analysis items: ADRs, etc.

Subgroup items: Sex [Male, Female]

Analysis method: Following analysis will be conducted for the above analysis items in each subgroup.

- (1)Number of patients with ADRs, etc.
- Number of incidence of ADRs, etc. (2)
- (3)Percentage of patients with ADRs, etc.
- Classification of ADRs, etc. (4)

The methods to count individual analysis items are the same as specified in

#### Section 4.2.2.

#### 4.4.3 Incidence of ADR/infection by age subgroup

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Age (year) Subgroup items:

[Min<= - <65, 65<= - <75, 75<= - <=Max] Certified the above analysis items in each ORs, etc Analysis method: Following analysis will be conducted for the above analysis items in each

subgroup.

- (1)Number of patients with ADRs, etc.
- (2)Number of incidence of ADRs, etc.
- Percentage of patients with ADRs, etc. (3)
- Classification of ADRs, etc. (4)

to the applica The methods to count individual analysis items are the same as specified in

Section 4.2.2.

# 4.4.4 Incidence of ADR/infection by purpose of NSAID therapy

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Purpose of NSAID therapy (multiple Subgroup items: [Rheumatoid arthritis, Osteoarthritis,

> counts) Others]

Analysis method: Following analysis will be conducted for the above analysis items in each

subgroup.

- Number of patients with ADRs, etc.
- (2)Number of incidence of ADRs, etc.
- (3)Percentage of patients with ADRs, etc.
- Classification of ADRs, etc. (4)

The methods to count individual analysis items are the same as specified in

Section 4.2.2.

#### 4.4.5 Incidence of ADR/infection by presence/absence of complication

Safety analysis set

Analysis items: ADRs, etc. Subgroup items: Existence of complication [Yes or No]

Analysis method: Following analysis will be conducted for the above analysis items in each subgroup.

- (1) Number of patients with ADRs, etc.
- (2) Number of incidence of ADRs, etc.
- (3) Percentage of patients with ADRs, etc.
- (4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in Section 4.2.2.

#### 4.4.6 Incidence of ADR/infection by presence/absence of renal disease

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Existence of renal disease [Yes or No]

Analysis method: Following analysis will be conducted for the above analysis items in each

subgroup.

(1) Number of patients with ADRs, etc.

- (2) Number of incidence of ADRs, etc.
- (3) Percentage of patients with ADRs, etc.
- (4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in Section 4.2.2.

# 4.4.7 Incidence of ADR/infection by presence/absence of hepatic disease

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Existence of hepatic disease [Yes or No]

Analysis method: Following analysis will be conducted for the above analysis items in each

subgroup.

(1) Number of patients with ADRs, etc.

(2) Number of incidence of ADRs, etc.

(3) Percentage of patients with ADRs, etc.

(4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in Section 4.2.2.

#### 4.4.8 Incidence of ADR/infection by BMI subgroup

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: BMI (kg/m<sup>2</sup>)

$$25.0 \le - \le Max$$

Analysis method: Following analysis will be conducted for the above analysis items in each

subgroup.

Number of patients with ADRs, etc. (1)

Number of incidence of ADRs, etc. (2)

(3)Percentage of patients with ADRs, etc.

(4)Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in

Section 4.2.2.

# 4.4.9 Incidence of ADR/infection by type of long-term NSAIDs

Safety analysis set Analysis

population:

Analysis items: ADRs, etc.

Type of long-term NSAIDs (at Subgroup items: [COX-2 inhibitors, Others]

the initial dose)

Analysis method: Following analysis will be conducted for the above analysis items in each Property of Takeda. For

subgroup.

(1)Number of patients with ADRs, etc.

(2)Number of incidence of ADRs, etc.

(3) Percentage of patients with ADRs, etc.

(4)Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in

Section 4.2.2.

# 4.4.10 Incidence of ADR/infection by presence/absence of concomitant drug (excluding NSAIDs)

Existence of concomitant drug (excluding [Yes or No] NSAIDs)

Analysis method: Following analysis will be conducted for the above analysis items in each subgroup.

(1) Number of patients with ADRs, etc.
(2) Number of incidence of ADRs, etc.
(3) Percentage of patients with ADRs, etc.
(4) Classification of ADRs, etc.
The methods to count individual analysis items are the same as Section 4.2.2.

only and subil

#### 4.4.11 Change of liver function test value

Analysis Safety analysis set

population:

AST (IU/L), ALT (IU/L), y-GTP (IU/L), ALP (IU/L), Total bilirubin (mg/dL), Analysis items:

LDH (IU/L), Serum gastrin (pg/mL)

Summary statistics will be calculated for the measured values of each Analysis method:

analysis items. In interval (two-sided) of me Tablets will be calculated. evaluation period [at the start of treatment, at the completion of survey] for the above analysis items. In addition, summary statistics and 95% confidence interval (two-sided) of mean change from the start of treatment with Takecab

#### 5 Tabulated analysis on efficacy results

# 5.1 Development of gastric ulcer, duodenal ulcer, or hemorrhagic lesions in stomach or duodenum

Analysis Efficacy analysis set

population:

Analysis items: Development of gastric ulcer, duodenal [Yes or No]

ulcer, or hemorrhagic lesions in stomach or

duodenum

Breakdown (multiple counts)

Development of gastric ulcer [Yes or No] Development of duodenal ulcer [Yes or No]

Development of hemorrhagic lesions in

[Yes or No

stomach

[Yes or No] Development of hemorrhagic lesions in

duodenum

Analysis method: Frequency will be counted for the above analysis items, and point estimates and

95% confidence interval (two-sided) of proportions of patients who developed

ulcer or hemorrhagic lesions will be calculated.

# 5.2 Development of gastric ulcer, duodenal ulcer, or hemorrhagic lesions in stomach or duodenum (count in each subgroup)

Efficacy analysis set Analysis

population:

Analysis items: Development of gastric ulcer, duodenal [Yes or No]

ulcer, or hemorrhagic lesions in stomach or

duodenum

Breakdown (multiple counts)

Development of gastric ulcer [Yes or No] Development of duodenal ulcer [Yes or No] Development of hemorrhagic lesions in [Yes or No]

Development of hemorrhagic lesions in [Yes or No]

duodenum

Property of Takeda. For Sex [Male, Female]

[Min<= - <65, 65<= - <75, Age (year)

 $75 \le - \le Max$ 

Existence of H. pylori infection [Positive or Negative or Unknown] BMI (kg/m<sup>2</sup>)

[Min<= - <18.5, 18.5<= - <25.0,

 $25.0 \le - \le Max$ 

Type of long-term NSAIDs (at the initial [COX-2 inhibitors,

dose) Others]

Terms of Use as, and anos of a sculated. Let a depart and a subject to the applicable only and a subject to the applicable only and a subject to the applicable only and a subject to the applicable only and a subject to the applicable of the applicable of the applicability o Analysis method: Frequency by each subgroup will be counted for the above analysis items, and

29

#### 6 Incidence of ADR/infection in additional pharmacovigilance activities

# Terms of Use Incidence of ADR/infection in additional pharmacovigilance activities (Attachment Form

12)

Analysis Safety analysis set

population:

Analysis items: ADRs, etc. falling under the category of safety specification (described as

important identified risks, important potential risks, and important missing

information)

Subgroup items: Seriousness [Serious, Non-serious]

Following analysis will be conducted for the above analysis items in each Analysis method:

subgroup in accordance with Notes 1 to 4 in Attachment Form 12 included in

PSEHB/PED Notification No. 1128-2 (reexamination notification) dated

November 28, 2017.

Number and proportion of patients with ADRs, etc. (1) Property of Takeda. For non-commercial use only and approperty of Takeda. Risk terms and their order of listing will follow those of important identified

risks, important potential risks, and important missing information.

#### Outline of patients in postmarketing surveillance, etc.

#### Outline of patients in postmarketing surveillance, etc. (Attachment Form 16)

Analysis

population:

Analysis items:

case name)

.case name)

Analysis method: A list will be prepared for the above analysis items in accordance with Notes 1 to

3 in Attachment Form 16 included in PSEHB/PED Notification No. 1128-2

Property of Takedai. For non-com (reexamination notification) dated November 28, 2017.

| Version | Date | Person who prepared/revised this document | Comment |
|---|---|---|---|
| Version 1 | 2020.11.9 | PPD | Preparation of Version 1 |

aim 1 ion 1